CLINICAL TRIAL: NCT04471701
Title: Italian Web-based EPICOVID19 Cross-sectional Survey
Brief Title: Italian Web-based Cross-sectional Survey on COVID-19
Acronym: EPICOVID19
Status: Completed | Type: Observational
Sponsor: Institute of Biomedical Technologies-National Research Council, Italy (Other)
Collaborators: National Research Council, Institute of Clinical Physiology, Italy (Other); Institute of Neuroscience-National Research Council (Unknown); University of Milan (Other); Italian Society of Gerontology and Geriatrics (Unknown); Italian Society for Infectious and Tropical Diseases (Unknown)
Responsible Party: Sponsor
Other Study IDs: EPICOVID19_2020
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-09

CONDITIONS: Covid19; SARS-CoV Infection; Survey, Family Life; Epidemic Disease; Self-Assessment
Keywords: SARS-CoV-2;COVID-19;voluntary respondents;web-based survey
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Environmental Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Environmental exposure and clinical features — Environmental exposures and clinical features are measured by means of a self-administered 38-item on-line questionnaire containing mainly mandatory and closed questions divided into six sections: i) socio-demographic data; ii) clinical evaluation; iii) personal characteristics and health status; iv) housing conditions; v) lifestyle; and vi) behaviours following the lockdown.

SUMMARY:
The outbreak of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) that started in late December 2019 in the Hubei province of China caused millions of cases worldwide in just a few months, and evolved into a real pandemic.

However, only approximately 20% of SARS-CoV-2 infected patients required intensive on sub-intensice medical care and the remained experience mild or subclinical form of the disease that did not require hospital admission and a relatively high percentage (40 to 45%) remained asymptomatic.

Understanding the occurrence of SARS-CoV-2-like infectious in a large non-hospitalized population, when the epidemic peak was occurring in Italy, is of paramount importance but data are scarce.

The goal of this research project is to estimate the number of suspected cases of COVID-19 and to investigate the role of the potential factors associated with SARS-CoV-2 infection in a large Italian sample of respondents living in Italy during the lockdown (started in Italy on 9 March 2020).

EPICOVID19 is an Italian countrywide self-administered cross-sectional web-based survey on adult volunteers launched on April 13, 2020.

The on-line questionnaire has been developed starting from the available literature and implemented using an open source platform focusing on beahvioural and clinical features of participants.

DETAILED DESCRIPTION:
The COVID-19 pandemic is posing an unprecedented threat worldwide, which have been experiencing widespread transmission of the virus in the community for several weeks.

During the epidemic peak, epidemiological surveillance strategies were mainly based on the testing of symptomatic patients with serious diseases requiring hospitalization and intensive or sub-intensive medical care. This has underestimated the real spread of the infection in the mild symptomatic (paucisymptomatic) or asymptomatic individuals or in specific group of persons with limited access to testing.

EPICOVID19 was developed and launched to accomplish the following objectives: i) to estimate the number of suspected cases of COVID-19 in the general population, and ii) to investigate the role of the potential factors associated with SARS-CoV-2 infection in adult volunteers living in Italy during the lockdown.

EPICOVID19 is a national Italian anonymous self-administered internet-based survey that was carried out using a cross-sectional research design in a convenience sample of adult volunteers (18+ years old) living in Italy during the lockdown. The survey was launched on 13 April 2020.

In order to enrol as many subjects as possible, the link to the electronic survey was uploaded, shared and disseminated via several channels: e-mails, social media platforms (Facebook, Twitter, Instagram, Whatsapp), press releases, internet pages, local radio and TV stations, and institutional websites that called upon volunteers to contact the study website https://epicovid19.itb.cnr.it/.

The EPICOVID19 study was established as a collaboration of a working work including epidemiologists, clinicians, biostatisticians, and public health professionals to improve SARS-CoV-2-related knowledge. The steering group tested the survey for a period of 2 weeks before starting to share the public link to the general population on April 13, 2020. The participants are asked to complete the self-administered 38-item questionnaire, which contained mainly mandatory and closed questions that is divided into six sections.

EPICOVID19 was designed by the steering group after a literature review of existing research into COVID-19. To guarantee the maximal comparability to other large epidemiological studies, several questions was chosen based on standardized and validated questionnaires. The survey was adapted to the national context and implemented using the European Commission's open-source official EUSurvey management tool (https://ec.europa.eu/eusurvey).

The survey includes an introductory page briefly describing the rational and the aims of the study, the consortium, and the option to provide or not the consent to participate.

The first section of the questionnaire investigates the socio-demographic characteristics of the respondents: sex at birth, birth year, ethnicity, user's postal code and municipality of residence, educational level, employment status, and current (or last) occupation.

The second section of the questionnaire investigates the clinical features: SARS-CoV-2 infection-like symptoms and the month of onset of the first symptoms, pre-existing diseases, other conditions to refer, vaccines, past and current use of medication and supplements, and, for females only, use of contraception or hormone replacement therapy at menopause, and number of completed pregnancies, when applicable. Data about close contact with confirmed or suspected cases, contacts with general practitioner and/or national emergency numbers, molecular tests and results (if available), hospitalization for confirmed or suspected SARS-CoV-2-like infection, and other possible risk conditions to refer, are also collected.

The third section of the questionnaire is focused on the personal characteristics and health status of respondents: questions about self-perceived health status and risk perception .

The fourth section investigates the housing conditions: population density in the area of residence, self-reported traffic intensity in the area of residence, number of rooms, number of co-habitants, and presence of at-risk co-habitants.

The fifth section focuses on lifestyles: daily mean number of contacts, smoking habit, and frequency of weekly physical activity.

The sixth section investigates the behaviours following the lockdown: job conditions, number of times of going out per week, and use of public transportation.

The Ethics Committee of the Istituto Nazionale per le Malattie Infettive I.R.C.C.S. Lazzaro Spallanzani (Protocol No. 70, 12/4/2020) approved the EPICOVID19 study protocol. When they first accessed the on-line platform, the participants were informed of the purpose of the study, the data to be collected, and the method of storage. The data were handled and stored in accordance with the European Union General Data Protection Regulation (EU GDPR) 2016/679 (http://gdpr-info.eu/), and data transfer was safeguarded by means of encrypting/decrypting and password protection. The study was conducted according to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* age of >=18 years;
* access to a mobile phone, computer, or tablet with internet connectivity;
* on-line consent to participate in the study.

Exclusion Criteria:

* age of <18 years;
* without access to a mobile phone, computer, or tablet with internet connectivity;
* not provide on-line consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: EPICOVID19 is a national Italian internet-based survey that targets adult volunteers (males and females >=18 years old) living in Italy during the lockdown (started in Italy on 9 March 2020). In order to enrol as many subjects as possible, the survey was promoted using social media (Facebook, Twitter, Instagram, Whatsapp), press releases, internet pages, local radio and TV stations, and institutional websites that called upon volunteers to contact the study website (https://epicovid19.itb.cnr.it/).
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants (%) with COVID-19-like symptoms | 3 months (July 2020) after initial data collection (April 2020)
  Measured by using answers on the Clinical evaluation section of the questionnaire: Fever > 37.5 °C for at least 3 consecutive days; cough; sore throat/rhinorrea; headache; myalgia; olfactory/taste disorders; shortness of breath; chest pain; tachycardia; gastrointestinal disorders; conjunctivitis.
  Variables on symptomatology will be created by considering each symtom singularly and by combining them using a priori definition (e.g. WHO) and a posteriori approach (based on EPICOVID19 data).
  Logistic regression models will be applied to assess the measurements of association between exposures of interest and COVID-19-like symptoms by estimating the aOR and 95%CI.
Number of participants (%) with SARS-CoV-2 nasopharyngeal swab (NPS) test positivity | 3 months (July 2020) after initial data collection (April 2020)
  Measured by using answers collected thorugh the on-line questionnaire about molecular NPS tests results.
  Logistic regression models will be applied to assess the measurements of association between exposures of interest and SARS-CoV-2 NPS positivity versus negativity by estimating the odds ratios (aOR) and 95% Confidence Intervals (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Federica Prinelli, PhD, Principal Investigator — Institute of Biomedical Technologies-National Research Council; Fulvio Adorni, MPH, Principal Investigator — Institute of Biomedical Technologies-National Research Council
Locations (1):
- Institute of Biomedical Technologies-National Research Council, Segrate, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prinelli F, Trevisan C, Noale M, Franchini M, Giacomelli A, Cori L, Jesuthasan N, Incalzi RA, Maggi S, Adorni F; EPICOVID19 Working Group. Sex- and gender-related differences linked to SARS-CoV-2 infection among the participants in the web-based EPICOVID19 survey: the hormonal hypothesis. Maturitas. 2022 Apr;158:61-69. doi: 10.1016/j.maturitas.2021.11.015. Epub 2021 Dec 4. PMID 35241240
- [Derived] Prinelli F, Bianchi F, Drago G, Ruggieri S, Sojic A, Jesuthasan N, Molinaro S, Bastiani L, Maggi S, Noale M, Galli M, Giacomelli A, Antonelli Incalzi R, Adorni F, Cibella F; EPICOVID19 Working Group. Association Between Smoking and SARS-CoV-2 Infection: Cross-sectional Study of the EPICOVID19 Internet-Based Survey. JMIR Public Health Surveill. 2021 Apr 28;7(4):e27091. doi: 10.2196/27091. PMID 33668011
- [Derived] Trevisan C, Noale M, Prinelli F, Maggi S, Sojic A, Di Bari M, Molinaro S, Bastiani L, Giacomelli A, Galli M, Adorni F, Antonelli Incalzi R, Pedone C; EPICOVID19 Working Group. Age-Related Changes in Clinical Presentation of Covid-19: the EPICOVID19 Web-Based Survey. Eur J Intern Med. 2021 Apr;86:41-47. doi: 10.1016/j.ejim.2021.01.028. Epub 2021 Jan 29. PMID 33579579
- [Derived] Adorni F, Prinelli F, Bianchi F, Giacomelli A, Pagani G, Bernacchia D, Rusconi S, Maggi S, Trevisan C, Noale M, Molinaro S, Bastiani L, Fortunato L, Jesuthasan N, Sojic A, Pettenati C, Tavio M, Andreoni M, Mastroianni C, Antonelli Incalzi R, Galli M. Self-Reported Symptoms of SARS-CoV-2 Infection in a Nonhospitalized Population in Italy: Cross-Sectional Study of the EPICOVID19 Web-Based Survey. JMIR Public Health Surveill. 2020 Sep 18;6(3):e21866. doi: 10.2196/21866. PMID 32650305
- See also: Institutional web-site of ITB-CNR — http://epicovid19.itb.cnr.it/
- See also: Rapid COVID-19 Screening Based on Self-Reported Symptoms: Psychometric Assessment and Validation of the EPICOVID19 Short Diagnostic Scale — https://www.jmir.org/2021/1/e23897/
- See also: Self-Reported Symptoms of SARS-CoV-2 Infection in a Nonhospitalized Population in Italy: Cross-Sectional Study of the EPICOVID19 Web-Based Survey — https://publichealth.jmir.org/2020/3/e21866/